CLINICAL TRIAL: NCT02564380
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of Pembrolizumab Maintenance Following First-Line Platinum Based Chemotherapy in Patients With Metastatic Squamous - Non-Small Cell Lung Cancer (sNSCLC)
Brief Title: Study of Pembrolizumab Maintenance Following First-Line Platinum Based Chemotherapy in Patients With Metastatic Squamous - Non-Small Cell Lung Cancer (sNSCLC)
Acronym: PRIMUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Since trial start in Jan. 2016 only 41 patients could be recruited until planned date of end of follow up period. Under consideration of this fact the recruitment of the planned 130 patients was not possible within a reasonable recruitment period.
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIO-TRK-0115
Record Dates: First submitted 2015-09-10; First posted 2015-09-30 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Pembrolizumab (Experimental): Pembrolizumab 200 mg every three weeks until disease progression (maximum 2 years)
  Interventions: Drug: Pembrolizumab
- Arm B: Placebo (Placebo Comparator): Placebo i.v. every three weeks until disease progression (maximum 2 years)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pembrolizumab
  Other Names: MK-3475
  Arms: Arm A: Pembrolizumab
Drug: Placebo
  Arms: Arm B: Placebo

SUMMARY:
A Phase II Randomized, Double-Blind, Placebo-Controlled Study of Pembrolizumab Maintenance Following First-Line Platinum Based Chemotherapy in Patients with Metastatic Squamous - Non-Small Cell Lung Cancer (sNSCLC).

DETAILED DESCRIPTION:
Patients with squamous non-small cell lung cancer and an ECOG of 0-1 who received a first-line therapy with Cis-/Carboplatin for at least 2 cycles that had at least Complete Response (CR) / Partial Response (PR) / Stable Disease (SD) according to Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 will be randomized either to Arm A Pembrolizumab or to Arm B Placebo for a maximum of 2 years or until progressive disease or unacceptable toxicity.

The aim is to investigate the efficacy of Pembrolizumab vs. placebo in terms of progression-free survival in patients with metastatic squamous, non-small cell lung cancer. Furthermore to evaluate tumor response, survival, tolerability and safety as well as quality of life of patients receiving Pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, age ≥ 18 years
2. Signed informed consent
3. Ability to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
5. At least one measurable tumor lesion according to RECIST 1.1
6. Histologically or cytologically confirmed diagnosis of stage IV (AJCC Version 7) squamous non-small cell lung carcinoma
7. Complete response, partial response or stable disease after at least 2 cycles of first-line chemotherapy with cisplatin or carboplatin
8. Last administration of platinum based first-line chemotherapy ≤ 5 +/- 1 week(s) prior first dose of study treatment
9. Tumor specimen before first-line chemotherapy available for immunohistochemistry (IHC) of PD-L1 at a central laboratory. Tumor specimen must be a tumor block not a pre-cut slide.
10. Adequate bone-marrow and organ function:

    * Absolute neutrophil count ≥ 1.5 x 10^9/L and
    * Thrombocytes ≥ 100 x 10^9/L and
    * Hemoglobin ≥ 9 g/dL
    * International Normalized Ratio (for blood clotting time) (INR) ≤ 1.5 and Partial Thromboplastin Time (PPT) ≤ 1.5 x upper limit during the last 7 days before therapy
    * Bilirubin < 1.5 x Upper Limit of Normal (ULN) and
    * Aspartate aminotransferase ((AST (GOT)) and Alanine aminotransferase ((ALT) (GPT)) < 3 x ULN (5 x ULN in case of liver metastases)
    * Creatinine ≤ 1.5 x upper limit or creatinine clearance ≥ 45 mL/min (after first line chemotherapy)
11. In female patients of childbearing potential (i.e. did not undergo surgical sterilization - hysterectomy, bilateral tubal ligation, or bilateral oophorectomy - and is not post-menopausal for at least 24 consecutive months), a negative pregnancy test at screening
12. Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use 2 adequate barrier methods of contraception during study treatment and for 120 days after last administration of study drug

Exclusion Criteria:

Patients with any of the following will not be eligible for the study:

1. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start. It is permissable that a patient is in the follow-up phase of any previous study.
2. Patient received systemic steroid therapy within three days prior to the first dose of study treatment or received any other form of immunosuppressive medication
3. History of allogeneic tissue/solid organ transplant
4. History of pneumonitis or interstitial lung disease that has required oral or i.v. steroids
5. Radiotherapy of target lesion ≤ 28 days prior first dose of study treatment
6. Major surgery ≤ 28 days prior first dose of study treatment
7. Minor surgery (e.g. venous catheter) ≤ 24 hours prior first dose of study treatment
8. Cardiovascular or cerebrovascular disease of clinical relevance: e.g. acute myocardial infarction or stroke during the last 6 months, unstable angina, relevant and unstable dysrhythmia (controlled Tachyarrhythmia absoluta (TAA) allowed).
9. Wound healing disorders, active ulcus ventriculi/duodenal ulcer, bone fracture
10. Known active Hepatitis B virus (HBV), Hepatitis C virus (HCV) or HIV infection
11. Has any other active infection requiring systemic therapy.
12. Patients with active tuberculosis
13. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
14. Female patient pregnant or breastfeeding, or expecting to conceive or father children during the study and through 120 days after last administration of study drug
15. Indications of a neurological or other disease, which may influence the feasibility of the study or may seriously disturb tolerability
16. A diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
17. Patient has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. [Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.]
18. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
19. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
20. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
21. Has known hypersensitivity to pembrolizumab or any of its insipients.
22. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 Arzneimittelgesetz (AMG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2020-05-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 35 months.
  progression-free survival according to RECIST 1.1

SECONDARY OUTCOMES:
overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 35 months.
  Efficacy measure
overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 35 months.
  Efficacy measure
PD-L1 expression in tumor samples | samples at baseline taken ; collection up to 35 months
  assessment of the prognostic value of PD-L1 expression in tumor samples obtained prior to study enrollment
Safety (adverse events graded according to US NCI Common terminology criteria for adverse events) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 35 months.
  Safety (intensity and incidence of adverse events, graded according to US NCI Common terminology criteria for adverse events (CTCAE) Version 4.03)
Functional Assessment of Cancer Therapy for patients with Lung cancer | every 6 weeks until EOT for approx. 7 months
  with the FACT-L questionnaire as part of the quality of life assessment
Lung Cancer Symptom Scale (LCSS) | every 6 weeks until EOT for approx. 7 months
  as part of the quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reck, PD Dr., Principal Investigator — LungenClinic Grosshansdorf
Locations (1):
- LungenClinic Grosshansdorf, Großhansdorf, Germany

REFERENCES:
- See also: Description: Working Group for Medical Oncology (AIO) from the German Cancer Society (DKG) — http://www.aio-portal.de